CLINICAL TRIAL: NCT00852423
Title: Safe and Efficacious Artemisinin-based Combination Treatments for African Pregnant Women With Malaria
Acronym: PREGACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: National Institute for Medical Research, Tanzania (Other Government); Kwame Nkrumah University of Science and Technology (Other); Centre Muraz (Other); Kamuzu University of Health Sciences (Other); Tropical Diseases Research Centre, Zambia (Other Government); Institute of Tropical Medicine(KIT), Amsterdam (Unknown); Liverpool School of Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITMP0308
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Malaria in Pregnancy
Keywords: Malaria in pregnancy; Sub-saharan Africa; Treatment; Artemisinin containing Therapy; Efficacy; Safety
MeSH Terms: interventions — amodiaquine, artesunate drug combination; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- DHAPQ (Experimental): Three-day treatment with dihydroartemisinin-piperaquine
  Interventions: Drug: Dihydroartemisinin-piperaquine
- MQAS (Experimental): Three-day treatment with mefloquine artesunate
  Interventions: Drug: Artesunate-mefloquine
- AQAS (Active Comparator): Three-day treatment with artesunate-amodiaquine
  Interventions: Drug: Artesunate-amodiaquine
- AL (Active Comparator): Three day treatment with artemether-lumefantrine (Coartem(R)
  Interventions: Drug: Artemether-lumefantrine

INTERVENTIONS:
Drug: Dihydroartemisinin-piperaquine — DHA-PQ tablets are green film coated intended for oral use and contain 20/160mg or 40/320mg of dihydroartemisinin (DHA) and piperaquine phosphate (PQ) respectively. In this trial the 40/320mg for adults will be used. Developed by Sigma Tau in partnership with Medicines for Malaria Venture.
  Other Names: DHAPQ, Eurartesim
  Arms: DHAPQ
Drug: Artesunate-mefloquine — MQAS will be provided as a fixed-dose ACT. There are 2 strengths (AS25+MQ55mg and AS100+MQ220mg) and dosing regimen is calculated according to 12 mg/kg AS and 24mg/kgMQ total dose over three days. Pregnant women will receive 2 tablets/day for 3 days. It is developed by Farmanguinhos with the Drugs for Neglected Diseases Initiative. To be noted: if the FDCs will not get the WHO pre-qualification before the start of recruitment, the separate AS and MQ will be used
  Other Names: MQAS
  Arms: MQAS
Drug: Artesunate-amodiaquine — AQAS, developed by teh DNDi with Sanofi-Aventis and manufactured by Sanofi-Aventis, has been pre-qualified by the WHO in 2008 and is available in several African countries, including those involved in this trial. AQ-AS tablets are round, yellow on one side and white-slightly yellow on the other, with a breaking bar, AS engraved on one side and either 25, 50 or 100 on the other side. Tablets to be used in this trial are those 100mg/270mg AS/AQ, containing 100 mg of artesunate, 352.640 mg of amodiaquine hydrochloride corresponding to 270mg of amodiaquine base.
  Other Names: AQAS, artesunate-amodiaquine Winthrop®
  Arms: AQAS
Drug: Artemether-lumefantrine — AL (tablets containing a FDC of 20 mg of artemether and 120 mg of lumefantrine) is manufactured by Novartis and has been extensively used in Africa for the treatment of uncomplicated malaria. AL was registered in Switzerland in 1999, has since received marketing authorisation in several endemic and non-endemic countries and it is WHO pre-qualified.
  Other Names: AL, Coartem, Riamet
  Arms: AL

SUMMARY:
Malaria is the most important human parasitic disease and is responsible of high morbidity and mortality in resource-poor countries. Pregnant women, who are a high-risk group, are almost always excluded from clinical trials; thus, the investigators lack sufficient information on the safety and efficacy of most antimalarials in pregnancy. The recommendation of the World Health Organization to use artemisinin combination therapy (ACT) in the 2nd and 3rd trimester is already implemented in several African countries, however documentation of their efficacy and safety in pregnancy is still limited. Thus, the investigators propose to evaluate the efficacy and safety of 4 ACT(artemether-lumefantrine, amodiaquine-artesunate, mefloquine-artesunate and dihydroartemisinin-piperaquine), when used to treat pregnant women with P. falciparum malaria; the results will help to recommend the optimal therapy for this high-risk group in Africa.

DETAILED DESCRIPTION:
Malaria is the most important human parasitic disease. Although pregnant women are a high-risk group, they are almost systematically excluded from clinical trials, for fear of teratogenicity and embryotoxicity; thus, we generally lack sufficient information on the safety and efficacy of most antimalarials in pregnancy, as well as evidence-based recommendations for the prevention and treatment of malaria during pregnancy.

The WHO recommendation to use artemisinin combination therapy (ACT) in the 2nd and 3rd trimester is already implemented in several African countries. However, the documentation of their efficacy and safety in pregnancy is still limited, especially concerning the African contexts.

Therefore, we propose to test 4 fixed-dose combinations (artemether-lumefantrine, amodiaquine-artesunate, mefloquine-artesunate and dihydroartemisinin-piperaquine), to evaluate their efficacy and safety when administered to pregnant women (2nd and 3rd trimester) infected with P. falciparum. Explanatory variables will be collected for treatment failure (PCR-corrected) and for recurrent parasitaemia. The primary hypothesis tested will be the clinical equivalence (pair-wise non-inferiority) of the 4 treatment regimens with clinical equivalence defined as difference in treatment failure rates (PCR corrected) of 5% or less.

In addition, an attempt will be done to carry out in vitro testing at the time of recurrent infection. However, the success of the test will depend on the parasite density. In addition, blood samples collected on filter paper at day 0 and at day of recurrent parasitaemia will be genotyped for the search of known molecular markers related to drug resistance. Not all samples will be analyzed; rather these will be selected according to the therapeutic response so that the prevalence of molecular markers will be compared between treatment successes, true treatment failures and new infections.

ELIGIBILITY:
Inclusion Criteria:

* Gestation of at least 16 weeks and <37 weeks;
* P. falciparum monoinfection of any density, with or without symptoms
* Hb equal or higher than 7 g/dL;
* At least 15 years old;
* Residence within the health facility catchment's area;
* Willing to deliver at the health facility;
* Willing to adhere to study requirements (including in Zambia and Malawi, HIV VCT)
* Ability to provide written informed consent; if the woman is minor of age/not emancipated, the consent must be given by a parent or legal guardian according to national law (however, in this case, the investigator is responsible to check that the woman herself is also freely willing to take part in the study, and the woman will be asked to sign for "assent").

Exclusion Criteria:

* History of allergic reactions to the study drugs;
* History of known pregnancy complications or bad obstetric history such as repeated stillbirths or eclampsia;
* History or presence of major illnesses likely to influence pregnancy outcome including diabetes mellitus, severe renal or heart disease, or active tuberculosis;
* Current cotrimoxazole prophylaxis or ARV treatment;
* Any significant illness at the time of screening that requires hospitalization, including severe malaria;
* Intent to move out of the study catchment area before delivery or deliver at relative's home out of the catchment area.
* Prior enrollment in the study or concurrent enrollment in another study.
* Unable to take oral medication
* Clear evidence of recent (1 week) treatment with antimalarials or antimicrobials with antimalarial activity (clindamycin; azythromycin; etc.)

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3428 (Actual)
Dates: Start 2010-06; Primary Completion 2013-10 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Treatment Failure (PCR adjusted) | Day 63
Safety profiles including significant changes in relevant laboratory values | Until delivery

SECONDARY OUTCOMES:
Time to failure | Case by case
PCR unadjusted treatment failure | Day 63
Gametocyte carriage (gametocyte-weeks) | Case by case
Asexual parasite clearance time | Days to 2 consecutive negative blood slides.
Gametocytaemia (prevalence and density) | Day 7, 14, 21, 28 and 63 after treatment
Haemoglobin changes | Days 14, 28, 42 and 63
The presence of acute, chronic or past infection of the placenta (prevalence) | Delivery
Mean birth weight and prevalence of low birth weight newborns | Delivery
In vitro vitro and search of molecular markers related to drug resistance | At the time of recurrent infection
Determination of the PK profile of MQ, AQ and PQ (on 120 women/treatment) | Case by case

CONTACTS AND LOCATIONS:
Overall Officials: Umberto D'Alessandro, MD, Study Chair — Institute Tropical Medicine Belgium and MRC Unit in The Gambia; Tinto Halidou, PharmD, Principal Investigator — Centre Muraz
Locations (7):
- Burkina Faso (2):
  - ISSR/Centre Muraz, Nanoro
  - ISSR/Centre Muraz, Nazoanga
- Ghana (3):
  - Kwame Nkrumah University of Science & Technology, Kumasi, Ejisu Sekyere East, Ashanti Region
  - Kwame Nrumah University of Science and Technology, Kumasi, Juaben Government Hospital, Ashanti Region
  - Effiduase Government Hospital, Effiduase
- College of Medicine, University of Malawi, Chikwawa District Hospital, Blantyre, Malawi
- St Paul Hospital, Nchelenge, Nchelenge District, Zambia

REFERENCES:
- [Result] PREGACT Study Group; Pekyi D, Ampromfi AA, Tinto H, Traore-Coulibaly M, Tahita MC, Valea I, Mwapasa V, Kalilani-Phiri L, Kalanda G, Madanitsa M, Ravinetto R, Mutabingwa T, Gbekor P, Tagbor H, Antwi G, Menten J, De Crop M, Claeys Y, Schurmans C, Van Overmeir C, Thriemer K, Van Geertruyden JP, D'Alessandro U, Nambozi M, Mulenga M, Hachizovu S, Kabuya JB, Mulenga J. Four Artemisinin-Based Treatments in African Pregnant Women with Malaria. N Engl J Med. 2016 Mar 10;374(10):913-27. doi: 10.1056/NEJMoa1508606. PMID 26962727
- [Derived] Patson N, Mukaka M, D'Alessandro U, Chapotera G, Mwapasa V, Mathanga D, Kazembe L, Laufer MK, Chirwa T. Joint modelling of multivariate longitudinal clinical laboratory safety outcomes, concomitant medication and clinical adverse events: application to artemisinin-based treatment during pregnancy clinical trial. BMC Med Res Methodol. 2021 Oct 9;21(1):208. doi: 10.1186/s12874-021-01412-9. PMID 34627141
- [Derived] Nambozi M, Tinto H, Mwapasa V, Tagbor H, Kabuya JB, Hachizovu S, Traore M, Valea I, Tahita MC, Ampofo G, Buyze J, Ravinetto R, Arango D, Thriemer K, Mulenga M, van Geertruyden JP, D'Alessandro U. Artemisinin-based combination therapy during pregnancy: outcome of pregnancy and infant mortality: a cohort study. Malar J. 2019 Mar 28;18(1):105. doi: 10.1186/s12936-019-2737-7. PMID 30922317
- [Derived] PREGACT Study Group; Pekyi D, Ampromfi AA, Tinto H, Traore-Coulibaly M, Tahita MC, Valea I, Mwapasa V, Kalilani-Phiri L, Kalanda G, Madanitsa M, Ravinetto R, Mutabingwa T, Gbekor P, Tagbor H, Antwi G, Menten J, De Crop M, Claeys Y, Schurmans C, Van Overmeir C, Thriemer K, Van Geertruyden JP, D'Alessandro U, Nambozi M, Mulenga M, Hachizovu S, Kabuya JB, Mulenga J. Four artemisinin-based treatments in African pregnant women with malaria. Malawi Med J. 2016 Sep;28(3):139-149. PMID 27895848
- [Derived] Tahita MC, Tinto H, Yarga S, Kazienga A, Traore Coulibaly M, Valea I, Van Overmeir C, Rosanas-Urgell A, Ouedraogo JB, Guiguemde RT, van Geertruyden JP, Erhart A, D'Alessandro U. Ex vivo anti-malarial drug susceptibility of Plasmodium falciparum isolates from pregnant women in an area of highly seasonal transmission in Burkina Faso. Malar J. 2015 Jun 20;14:251. doi: 10.1186/s12936-015-0769-1. PMID 26088768
- [Derived] Nambozi M, Mulenga M, Halidou T, Tagbor H, Mwapasa V, Phiri LK, Kalanda G, Valea I, Traore M, Mwakazanga D, Claeys Y, Schurmans C, De Crop M, Menten J, Ravinetto R, Thriemer K, Van Geertruyden JP, Mutabingwa T, D'Alessandro U; Pregact Group. Safe and efficacious artemisinin-based combination treatments for African pregnant women with malaria: a multicentre randomized control trial. Reprod Health. 2015 Jan 15;12:5. doi: 10.1186/1742-4755-12-5. PMID 25592254